CLINICAL TRIAL: NCT00858351
Title: A Placebo-Controlled Trial of Thermal Biofeedback Assisted Relaxation for the Treatment of Diabetic Neuropathy: An Evaluation of Outcomes and Mechanisms
Brief Title: Thermal Biofeedback for the Treatment of Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Insulin Dependent Diabetes Trust (Unknown); American Pain Society (Other); Rosalind Franklin University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Angela Fidler Pfammatter, PhD, Postdoctoral Fellow, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200.97PY
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: Diabetes; Neuropathy; Peripheral; Painful; Thermal; Temperature; Biofeedback; Relaxation; Diabetic
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thermal Biofeedback Assisted Relaxation (Experimental)
  Interventions: Behavioral: Thermal Biofeedback Assisted Relaxation
- Discussion (Active Comparator)
  Interventions: Behavioral: Discussion with therapist

INTERVENTIONS:
Behavioral: Thermal Biofeedback Assisted Relaxation — 6 sessions, 25 minutes in duration of relaxation and imagery training while temperature of hands and feet are recorded.
  Arms: Thermal Biofeedback Assisted Relaxation
Behavioral: Discussion with therapist — 6 sessions, 25 minutes each, discussing topics with a therapist.
  Arms: Discussion

SUMMARY:
The purpose of this study is to examine potential treatment options for a condition in diabetics that causes tingling, pain, and numbness in the hands and /or feet, also known as diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Participants attend 6 sessions lasting from 35 minutes to 2 hours (depending on the session). Sessions can be scheduled once or twice per week. Sessions involve a walking task, filling out questionnaires, and having temperature of hands and feet monitored. This study involves no drugs, blood draws, or any other invasive procedures. Participants are urged to continue the treatment of diabetes and diabetic neuropathy as directed by their physician for the duration of their involvement with the study. After 3 months, a packet of questionnaires will be mailed with a stamped addressed envelope to be returned.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Diabetic Neuropathy in Hands and/or Feet
* Must have some sensation left in hands and feet

Exclusion Criteria:

* Any partial or total amputation of an limb or digit
* Any previous experience with biofeedback
* Prior treatment for alcohol abuse
* Severe Psychopathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-11; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Subjective Pain | Change in subjective pain rating from baseline to end of intervention

SECONDARY OUTCOMES:
Perceived Control | Change from mid-intervention (visit 4) to end of intervention
Temperature | Change within each session and across sessions from baseline to end of intervention